CLINICAL TRIAL: NCT05860257
Title: Transforming Adolescent Mental Health Through Accessible, Scalable, Technology-supported Small-group Instruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Arizona State University (Other); University of Wisconsin, Madison (Other); Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000719
Record Dates: First submitted 2023-03-20; First posted 2023-05-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Depression; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Investigators will allocate 20 high schools to intervention vs. control groups. Investigators will recruit in two cohorts (Fall 2023 and Fall 2024). Students will be in 9th grade in the first year, and will be followed into 10th, 11th, and then 12th grade, so in total the investigators will be working in each school for four years.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation of PeerLearning.net (Experimental): Teachers in implementation schools will be given access to training and resources to implement PeerLearning.net as a core component of instruction. Investigators will not create specific requirements of teachers but will ask that they deliver lessons with PeerLearning.net at least four times per month. Investigators will monitor all teacher usage and thus will be able to promote greater usage by (1) publicly acknowledging teachers that are using it frequently and experiencing success, and (2) targeting teachers who use it infrequently with additional resources and support to encourage more frequent use.
  Interventions: Behavioral: PeerLearning.net
- Pre-Intervention (No Intervention): Teachers in pre-intervention schools will continue with business as usual (i.e., typical instruction). Based upon previous experience in conducting research in school settings, teachers in pre-intervention schools will likely use CL very infrequently, and without the benefit of technology support.

INTERVENTIONS:
Behavioral: PeerLearning.net — PeerLearning.net provides an easy-to-use, scalable, and widely accessible means to support teachers in effectively designing and delivering high-fidelity Cooperative Learning (CL) lessons and, in turn, it has the potential to amplify the positive effects of CL found in previous research. Using PeerLearning.net, teachers design their lesson by selecting from among a set of typical CL lesson templates (e.g., jigsaw, peer tutoring, group projects) which they can customize and populate with their own curriculum and materials. These design templates represent the optimal, high-fidelity design that is required in order for CL to be successful. During lesson delivery, PeerLearning.net manages membership in learning groups, distributes instructional materials, directs student activities according to a pre-specified timetable, supports teacher observations of student behavior, and delivers post-lesson group activities and reviews.
  Arms: Implementation of PeerLearning.net

SUMMARY:
Adolescence is a developmental period of significant risk for anxiety, depressive symptoms, and suicidality, and the investigators propose to target key peer-based risk and protective factors using Cooperative Learning (CL). CL is a small-group instructional approach that can enhance peer relations and reduce peer-related risks, as well as promote academic engagement and achievement and reduce racial disparities. CL will be delivered with the aid of technology that automates the design and delivery of CL lessons, promoting rapid implementation, scalability, high fidelity, accessibility, and sustainability.

DETAILED DESCRIPTION:
Internalizing symptoms (i.e., anxiety, depressive symptoms, suicidality) are alarmingly common among adolescents. In 2019, nearly 37% of high school students reported feeling anxious, sad, or hopeless, representing an increase from 2017 (i.e., 31%), and nearly 19% seriously considered suicide, an increase from 2017 (17%). The coronavirus pandemic has exacerbated this problem, with research finding that social isolation resulting from the pandemic was linked to higher levels of stress, fear, loneliness, anxiety, depression, and suicide ideation among adolescents. Importantly, ethnic/racial disparities have been documented in internalizing symptoms, with more negative outcomes for Latinas and Black males. Current universal school-based approaches to prevention have reported uneven or limited effects, or no effects at all. Questions have also been raised regarding cost and accessibility. Despite the uneven track record of universal school-based (Tier 1) approaches, which has led some to recommend an emphasis on targeted (Tier 2) approaches, Tier 1 programs possess several advantages. First, given the demographic heterogeneity in risk factors, as well as disparate access to high-quality, culturally-sensitive health care, schools remain attractive as Tier 1 programs can ensure equitable access to primary prevention services. Second, universal programs avoid the difficulty of identifying adolescents at risk, and third, Tier 1 programs minimize the risk of stigmatizing adolescents who seek out or are referred to services. In this project, submitted to the Transformative Research Award initiative, the investigators will use cooperative learning (CL) as a universal (Tier 1) school-based prevention program to target malleable peer-based risk factors and subsequently evaluate how change in these mechanisms can reduce adolescent internalizing symptoms. CL targets various forms of maladaptive peer relations that create stress and comprise a significant risk factor for internalizing symptoms in adolescence; CL also promotes peer protective factors that can reduce the likelihood of internalizing symptoms (e.g., peer acceptance). CL has also been found to promote more cross-race interaction and interracial attraction, greater cross-ethnic academic support, and more frequent cross-ethnic friendships. To support teachers in implementing CL, the investigators will use a Web-based software platform that provides an accessible, high-fidelity mechanism to deliver CL lessons. The investigators will not only test for intervention effects, but will also evaluate the relative strength of specific, theoretically-derived change mechanisms, and uncover key issues/barriers related to implementation that will allow the investigators to dynamically adjust our implementation approach to achieve maximum impact during subsequent scale-up. This project is designed to establish feasibility with teachers and schools and counter potential threats to implementation fidelity while also creating a roadmap to enhanced scalability and sustained implementation. Significant results from this project could inspire broad uptake of this approach in educational contexts, potentially addressing a significant public health need during a time of crisis due to the coronavirus pandemic.

ELIGIBILITY:
Inclusion Criteria:

* All students and teachers in target grades in participating schools.

Exclusion Criteria:

* None.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7 | Fall of Year 1
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Spring of Year 1
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Fall of Year 2
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Spring of Year 2
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Fall of Year 3
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Spring of Year 3
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Fall of Year 4
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Generalized Anxiety Disorder 7 | Spring of Year 4
  Anxiety (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Fall of Year 1
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Spring of Year 1
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Fall of Year 2
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Spring of Year 2
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Fall of Year 3
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Spring of Year 3
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Fall of Year 4
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Patient Health Questionnaire | Spring of Year 4
  Depressive symptoms (scores zero to 3, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Fall of Year 1
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Spring of Year 1
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Fall of Year 2
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Spring of Year 2
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Fall of Year 3
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Spring of Year 3
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Fall of Year 4
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Youth Risk and Behavior Survey | Spring of Year 4
  Suicide ideation (scores zero to 6, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Fall of Year 1
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Spring of Year 1
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Fall of Year 2
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Spring of Year 2
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Fall of Year 3
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Spring of Year 3
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Fall of Year 4
  Service utilization (scores zero to 20, higher scores imply worse outcome)
Service Assessment for Children and Adolescents | Spring of Year 4
  Service utilization (scores zero to 20, higher scores imply worse outcome)

SECONDARY OUTCOMES:
Everyday Discrimination Scale | Fall of Year 1
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Spring of Year 1
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Fall of Year 2
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Spring of Year 2
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Fall of Year 3
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Spring of Year 3
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Fall of Year 4
  Discrimination (scores zero to 4, higher scores imply worse outcome)
Everyday Discrimination Scale | Spring of Year 4
  Discrimination (scores zero to 4, higher scores imply worse outcome)
University of Illinois Bully Scale | Fall of Year 1
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Spring of Year 1
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Fall of Year 2
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Spring of Year 2
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Fall of Year 3
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Spring of Year 3
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Fall of Year 4
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
University of Illinois Bully Scale | Spring of Year 4
  Bullying and victimization (scores 1 to 5, higher scores imply worse outcome)
Child Peer Social Skills Scale | Fall of Year 1
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Spring of Year 1
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Fall of Year 2
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Spring of Year 2
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Fall of Year 3
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Spring of Year 3
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Fall of Year 4
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Child Peer Social Skills Scale | Spring of Year 4
  Peer acceptance (scores 1 to 5, higher scores imply better outcome)
Perceived Stress Scale | Fall of Year 1
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Spring of Year 1
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Fall of Year 2
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Spring of Year 2
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Fall of Year 3
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Spring of Year 3
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Fall of Year 4
  Stress (scores 0 to 4, higher scores imply worse outcome)
Perceived Stress Scale | Spring of Year 4
  Stress (scores 0 to 4, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Fall of Year 1
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Spring of Year 1
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Fall of Year 2
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Spring of Year 2
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Fall of Year 3
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Spring of Year 3
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Fall of Year 4
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Adolescent Stress Questionnaire | Spring of Year 4
  Social stress (scores 1 to 5, higher scores imply worse outcome)
Classroom Life Scale | Fall of Year 1
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Spring of Year 1
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Fall of Year 2
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Spring of Year 2
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Fall of Year 3
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Spring of Year 3
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Fall of Year 4
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
Classroom Life Scale | Spring of Year 4
  Peer academic support (scores 1 to 5, higher scores imply better outcome)
School Attendance | Fall of Year 1
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Spring of Year 1
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Fall of Year 2
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Spring of Year 2
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Fall of Year 3
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Spring of Year 3
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Fall of Year 4
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
School Attendance | Spring of Year 4
  Degree of truancy (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Fall of Year 1
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Spring of Year 1
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Fall of Year 2
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Spring of Year 2
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Fall of Year 3
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Spring of Year 3
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Fall of Year 4
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
Reasons for Non-Attendance | Spring of Year 4
  Social issues causing non-attendance (scores 0 to 4, lower scores imply better outcome)
UCLA Loneliness Scale | Fall of Year 1
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Spring of Year 1
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Fall of Year 2
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Spring of Year 2
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Fall of Year 3
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Spring of Year 3
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Fall of Year 4
  Loneliness (scores 1 to 3, lower scores imply better outcome)
UCLA Loneliness Scale | Spring of Year 4
  Loneliness (scores 1 to 3, lower scores imply better outcome)
Secondary School Readiness Inventory | Fall of Year 1
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Spring of Year 1
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Fall of Year 2
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Spring of Year 2
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Fall of Year 3
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Spring of Year 3
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Fall of Year 4
  School engagement (scores 1 to 5, higher scores imply better outcome)
Secondary School Readiness Inventory | Spring of Year 4
  School engagement (scores 1 to 5, higher scores imply better outcome)
Substance use | Fall of Year 1
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Spring of Year 1
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Fall of Year 2
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Spring of Year 2
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Fall of Year 3
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Spring of Year 3
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Fall of Year 4
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)
Substance use | Spring of Year 4
  Use of tobacco, alcohol, and marijuana (scores 1 to 5, lower scores imply better outcome)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arizona State University, Tempe, Arizona
  - U of Oregon, Eugene, Oregon
  - U of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Investigators will ensure that project data is submitted according to the NIH Data Sharing Regimen (i.e., descriptive/raw data will be submitted semi-annually, and submission of all other data will occur at the time of publication, or prior to the end of the grant, whichever occurs first). Consent forms will reflect this submission of data to be shared. Investigators will store study data as Excel datasets. Research staff will document the study protocol and datasets on a publicly accessible website that will include surveys, names and labels for all variables and values, and calculations for composite scores. Investigators will remove personal identifiers from datasets and replace them with randomly assigned identifiers.
Supporting Information: ICF
Time Frame: As noted above, descriptive/raw data will be submitted semi-annually, and submission of all other data will occur at the time of publication, or prior to the end of the grant, whichever occurs first.
Access Criteria: There is no criteria.